CLINICAL TRIAL: NCT03238105
Title: Treatment of Periorbicular Hyperchromia Comparing 10% Thioglycolic Acid Peeling Versus Pulsed Intense Light: a Randomized Trial
Brief Title: Treatment of Periorbicular Hyperchromia Comparing 10% Thioglycolic Acid Peeling Versus Pulsed Intense Light
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 48653215.5.0000.5327
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Periorbital Disorder
Keywords: Dark circles; Periorbital hyperchromia; Facial aesthetics
MeSH Terms: interventions — 2-mercaptoacetate; Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: The selected patients will have each region of periorbital hyperchromia (right and left) randomized to one of the treatments (split face study).
Who Masked: Outcomes Assessor
Masking Description: There will be 2 blinded evaluators who will not know which side of the periorbital hyperchromia (right or left) received which treatment (IPL or peeling of 10% thioglycolic acid). They will do the evaluation through photographs, comparing the photos before the treatments with the photos after 1, 2 and 3 sessions after the treatments, without knowing what therapeutic modality was adopted in each periorbital region.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intense pulsed light (Experimental): The application model will be 3 months of treatment with monthly interval between sessions, totaling 3 sessions. The parameters are as follows: frequency 15 J / cm2, pulse duration 15 ms, 1-2 passed as erythema. Eye protection for IPL will be used during all sessions.
  Interventions: Device: Intense Pulsed Light
- Peeling of 10% thioglycolic acid (Experimental): In the first session the acid will be applied for three minutes, and with each new session the duration time with the product will increase in three minutes, so that in the last session the duration of the application will be 9 minutes. For the application of the product will be used flexible cotton rod, sparing the region just below the eyelids of the lower eyelid 0.5cm, therefore, no other measure is necessary for eye protection. After the given time, the substance will be removed with lint with 0.9% saline solution.
  Interventions: Drug: Thioglycolic Acid

INTERVENTIONS:
Drug: Thioglycolic Acid — Monthly sessions for 3 months with progressive increase of the duration of contact time of the drug with the skin, 3, 6 and 9 minutes.
  Arms: Peeling of 10% thioglycolic acid
Device: Intense Pulsed Light — Monthly sessions for 3 months.
  Other Names: IPL
  Arms: Intense pulsed light

SUMMARY:
Periorbital hyperchromia (POH) or periorbital hyperpigmentation, commonly known as "dark circles", is a relatively common condition and a frequent reason for dermatological consultation. It is defined as brown-colored pigmentation, ranging from light to dark, which mainly involves the lower eyelids. POH affects individuals over a wide age range, including both sexes and all ethnicities, and is associated with a tired and aged facial appearance. The most commonly affected people are those with the highest skin phototypes. Although the prevalence is similar between sexes and age groups, POH is a more frequent complaint in women. The dark circles characteristic of POH can negatively impact patients' quality of life, although it is not a condition associated with morbidity. Despite its high prevalence, only a few well-designed studies were done to evaluate its therapeutic options. The intense pulsed light (IPL) and the thioglycolic acid are safe treatment options and promote the improvement of dark circles, but it is not known if one treatment differs from the other in relation to efficacy and adverse effects.

DETAILED DESCRIPTION:
It is a blinded randomized clinical trial, with the sample size calculated of 29 subjects, already considering 10% of possible losses and refusals. For this number was considered 80% power and significance level of 5%.

Selected patients will be invited to participate and informed about the characteristics of the study. If they do, they must sign a free and informed consent form.

At the first visit, some demographic data will be collected, including sex, age, phototype, history of smoking and / or alcohol consumption, family history of periocular hyperpigmentation, personal or family history of allergies and hours of sleep, for instance.Photographic registration will be done in a standardized way. After completion of the study, the photographs will be evaluated blindly by two evaluators, and they will not know before what therapeutic modality was adopted in each periorbital region. Clinical evaluation will be obtained through the application of the Global Aesthetic Improvement Scale (with the following grades: much better, better, better, no change, worse) and visual analogue scale for clinical improvement from 0 (no improvement) to 10 (complete improvement), both with monthly evaluations. Each patient will be submitted to the two proposed therapies, being a therapeutic procedure in the right periocular region and another in the left periocular region. Each periocular region will be randomized using the random.org program for treatment with 10% thioglycolic acid peeling or IPL. Both therapies will be performed at the same time in the monthly visits, totaling 3 months of treatment (3 sessions of IPL and 3 sessions of thioglycolic acid). The first visit will be for collection of demographic data, physical examination record, colorimetry and questionnaire completion. Visits 2, 3 and 4 will be for the treatments and the visit in month 5 will be for evaluation of the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periocular hyperchromia diagnosed by clinical examination. The volunteers included must have a pigmentary component, which may or may not present the anatomical component, determined through physical examination with the aid of dermoscopy, to be performed at the inclusion study visit.

Exclusion Criteria:

* Pregnant patients, active collagenase patients, patients using photosensitizing substances and areas with bacterial or viral infections, patients with scars or tattoos at the evaluated site, patients undergoing any treatment modality for periocular hyperpigmentation in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response and compare treatment results | 5 months
  Through photographs the blinded evaluators will classify the difference on each side (right or left) using the Global Aesthetic Improvement (GAIS) scale. The evaluation will be comparing photographs before treatment with photographs after treatment. The data will be compared between the 2 treatments to evaluate if there was difference between them.

SECONDARY OUTCOMES:
Quality of Life Index in Dermatology | 5 months
  To evaluate the impact of periocular hyperpigmentation on patients' dermatological quality of life before and after treatments.
Pittsburgh Sleep Quality Index | at 1 day visit 1
  To evaluate the sleep quality on patients with periocular hyperpigmentation.
Adverse effects | 5 months
  To evaluate the immediate, early and late adverse effects related to the proposed treatments through questionnaires after each session and before the next session

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Boza, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided